CLINICAL TRIAL: NCT03031496
Title: An Open-label, Randomized, Single-dose, Two-period Cross-over Study to Evaluate Bioequivalence of GSK3542503 Hydrochlorothiazide + Amiloride Hydrochloride 50 mg: 5 mg Fixed Dose Combination Tablets Versus Reference Product in Healthy Adult Participants Under Fasting Conditions
Brief Title: Bioequivalence Study Between GSK3542503 Hydrochlorothiazide + Amiloride Hydrochloride 50 mg: 5 mg Tablets and Reference Product in Healthy Adult Participants Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 205694
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Hypertension
Keywords: Cross-over; Hydrochlorothiazide; Amiloride hydrochloride; Phase I; GSK3542503; Bioequivalence; FTIH
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide; Amiloride; amiloride, hydrochlorothiazide drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test A followed by Ref B of HCTZ 50mg+ Amiloride HCl 5mg (Experimental): Eligible participants following an overnight fast of at least 10 hours, will be administered the study drug orally with 240 mL (8 fluid ounces) of water. No food will be allowed for at least 4 hours post-dose. Water will be allowed as desired except for one hour before and after drug administration.
  Interventions: Drug: GSK3542503 (HCTZ 50mg/Amiloride HCl 5mg tablets); Drug: Moduretic (HCTZ 50mg/Amiloride HCl 5mg tablets)
- Ref B followed by test A of HCTZ 50mg + Amiloride HCl 5mg (Experimental): Eligible participants following an overnight fast of at least 10 hours, will be administered the study drug orally with 240 mL (8 fluid ounces) of water. No food will be allowed for at least 4 hours post-dose. Water will be allowed as desired except for one hour before and after drug administration.
  Interventions: Drug: GSK3542503 (HCTZ 50mg/Amiloride HCl 5mg tablets); Drug: Moduretic (HCTZ 50mg/Amiloride HCl 5mg tablets)

INTERVENTIONS:
Drug: GSK3542503 (HCTZ 50mg/Amiloride HCl 5mg tablets) — GSK3542503 (HCTZ 50mg/Amiloride HCl 5mg tablets) are cream-colored, circular, flat faced uncoated tablets with beveled edges having break line on one side and "BD" embossed on the other side.
Drug: Moduretic (HCTZ 50mg/Amiloride HCl 5mg tablets) — Moduretic (HCTZ 50mg/Amiloride HCl 5mg tablets) tablets are peach-colored, half scored, diamond shaped tablets marked "MSD917".

SUMMARY:
The combination of the diuretics amiloride hydrochloride (HCl) and hydrochlorothiazide (HCTZ) (GSK3542503) is indicated for the treatment of hypertension, congestive heart failure and hepatic cirrhosis with ascites and edema. This first time in human (FTIH) study is aimed to determine whether the test product GSK3542503 is bioequivalent to the reference (ref) hydrochlorothiazide 50 milligram (mg)/amiloride hydrochlorothiazide 5 mg in healthy adult participants under fasting conditions based on pharmacokinetic (PK) endpoints. This is a phase I, open label, balanced, randomized, single dose, two-way crossover study, enroling approximately 42 healthy participants at a single center. Study participants will be randomized to one of two treatment sequences (A-B or B-A) in accordance with the randomization schedule. A single dose of one of the two treatments A (Test: GSK3542503, a hydrochlorothiazide 50 mg and amiloride hydrochloride 5 mg fixed dose combination) or B (Reference: Moduretic, a hydrochlorothiazide 50 mg and amiloride hydrochloride 5 mg fixed dose combination), will be administered on Day 1, in each treatment period. Each participant will participate in both treatment periods and receive a single dose of each treatment. The treatment periods will be separated by a washout period of at least 7 days and no more than 14 days. The total duration in the study for each participant is expected to be 5 to 7 weeks, from screening to his or her last visit. A maximum of 42 participants will be randomized such that at least 32 evaluable participants complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy, non-smoker, as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* A participant with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the normal reference range for the population being studied may be included only if the investigator in consultation with the medical monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 19-30 kg/meter^2(inclusive).
* Healthy male or female participants

  * Male participants must agree to use contraception for 3 days after each dose of study treatment and refrain from donating sperm during that period.
  * A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: not a woman of childbearing potential (WOCBP), or a WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days after the last dose of study treatment.

The investigator is responsible for ensuring that male and female study participants understand how to correctly use the methods of contraception.

- Capable of giving signed informed consent, which includes compliance with the requirements and restrictions.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Abnormal renal function measured by creatinine clearance.
* Presence of hyperkalemia where the serum potassium is greater than upper limit of normal (ULN).
* History or known acute angle closure glaucoma or ocular complaints, which could increase the risk of ophthalmic reactions as deemed by the investigator.
* Abnormal BP as determined by the investigator.
* Alanine transaminase (ALT) >1.5 times ULN.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percentage).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Bazett's formula (QTcB) >450 milliseconds (msec). For purposes of data analysis, only QTcB, will be used.
* Past or intended use of over-the-counter or prescription medication including herbal medications, within 14 days prior to dosing. Specific medications listed in protocol of this study may be allowed.
* Where participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 90 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation within the last 90 days before signing of consent in this or any other clinical study involving an investigational study treatment.
* Presence of hepatitis B surface antigen (HBsAg) at screening, or a positive hepatitis C antibody test result at screening. Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative hepatitis C ribonucleic acid (RNA) test is obtained.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse.
* Sensitivity to heparin or heparin-induced thrombocytopenia.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy including allergy to penicillin and sulfonamides that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >21 units for males or > 14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Participants with any risk as defined in protocol of this study should be excluded from participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bloemfontein, South Africa

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20806

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a Phase I, open label, balanced, randomized, single dose, two-way crossover study, enrolling 42 healthy participants at a single center in South Africa.
Pre-assignment Details: Total 42 participants were enrolled and randomized to receive a single oral dose of study treatment in a cross-over manner.
Groups:
- Treatment A Followed by Treatment B: Eligible participants received a single oral dose of GSK3542503 (BIDURET), hydrochlorothiazide 50 milligrams (mg) and amiloride hydrochloride 5 mg fixed dose combination in Treatment Period 1. It was followed by a wash out period of 7 to 14 days. Participants received a hydrochlorothiazide 50 mg and amiloride hydrochloride 5 mg fixed dose combination in Treatment Period 2
- Treatment B Followed by Treatment A: Eligible participants received a single dose of moduretic, hydrochlorothiazide 50 mg and amiloride hydrochloride 5 mg fixed dose combination in Treatment Period 1. It was followed by a wash out period of 7 to 14 days. Participants received a single oral dose of GSK3542503 (BIDURET), hydrochlorothiazide 50 milligrams (mg) and amiloride hydrochloride 5 mg fixed dose combination in Treatment Period 2.
Period: Period 1
Arm/Group | Treatment A Followed by Treatment B | Treatment B Followed by Treatment A
Started | 21 | 21
Completed | 19 | 19
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2
Period: Period 2
Arm/Group | Treatment A Followed by Treatment B | Treatment B Followed by Treatment A
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Participants received a single oral dose of hydrochlorothiazide 50 milligrams (mg) and amiloride hydrochloride 5 mg fixed dose combination (either test or reference product) in each of the two treatment periods, separated by a wash out period of seven calendar days.
Arm/Group | All Subjects
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.1 (4.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American Heritage | 29
  White Heritage | 12
  Mixed Heritage | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) From Time Zero to the Time of the Last Quantifiable Concentration (AUC [0-t]) of Hydrochlorothiazide and Amiloride Hydrochloride
Description: Blood samples were collected at indicated time points under fasting conditions for pharmacokinetic (PK) analysis of hydrochlorothiazide and amiloride. Bioequivalence of test product and reference product was assessed based on the 90 percent confidence intervals (CIs) for estimates of the geometric mean ratios between the AUC (0-t) of the test and reference products in relation to the conventional bioequivalence range. An analysis of variance was used with sequence, subject (sequence), treatment and period as fixed effects.
Time Frame: Pre-dose, 0.33, 0.67, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10, 12,14, 16 hours post-dose on Day 1, 24 and 36 hours post dose on Day 2 and 48 hours post-dose on Day 3
Population: PK Population comprised of All participants who completed the study and for whom primary PK parameters was calculated for all treatment periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour x nanograms/milliliter (h*ng/mL)
Groups:
- Treatment A: Participants received a single oral dose of hydrochlorothiazide 50 milligrams (mg) and amiloride hydrochloride 5 mg fixed dose combination test product in each of the two treatment periods.
- Treatment B: Participants received a single oral dose of hydrochlorothiazide 50 milligrams (mg) and amiloride hydrochloride 5 mg fixed dose combination reference product in each of the two treatment periods
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 38 | 38
Hour x nanograms/milliliter (h*ng/mL)
  Hydrochlorothiazide | 2160 (22.0) | 2360 (18.8)
  Amiloride | 96.3 (22.9) | 94.1 (20.9)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — Bioequivalence of hydrochlorothiazide and amiloride hydrochloride was determined; Least square mean ratio = 91.52, 90% CI 2-sided [87.77 to 95.43] — Comparison of AUC (0-t) of hydrochlorothiazide for test and reference product has been presented
Statistical Analysis 2: Comparison: Treatment A vs Treatment B; Test type: Equivalence — Bioequivalence of hydrochlorothiazide and amiloride hydrochloride was determined; Least square mean ratio = 102.42, 90% CI 2-sided [98.12 to 106.91] — Comparison of AUC (0-t) of amiloride for test and reference product has been presented

2. Primary Outcome: Maximum Observed Concentration (Cmax) of Hydrochlorothiazide and Amiloride Hydrochloride in Plasma
Description: Blood samples were collected at indicated time points under fasting conditions for pharmacokinetic (PK) analysis of hydrochlorothiazide and amiloride. Bioequivalence of test product and reference product was assessed based on the 90 percent CIs for estimates of the geometric mean ratios between the Cmax of the test and reference products in relation to the conventional bioequivalence range. An analysis of variance was used with sequence, subject (sequence), treatment and period as fixed effects.
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 38 | 38
ng/mL
  Hydrochlorothiazide | 312 (28.5) | 377 (23.4)
  Amiloride | 9.27 (26.8) | 8.92 (25.4)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — Bioequivalence of hydrochlorothiazide and amiloride hydrochloride was determined; Least square mean ratio = 82.86, 90% CI 2-sided [77.37 to 88.74] — Comparison of Cmax of hydrochlorothiazide for test and reference product has been presented
Statistical Analysis 2: Comparison: Treatment A vs Treatment B; Test type: Equivalence — Bioequivalence of hydrochlorothiazide and amiloride hydrochloride was determined; Least square mean ratio = 103.92, 90% CI 2-sided [97.42 to 110.86] — Comparison of Cmax of amiloride for test and reference product has been presented

3. Secondary Outcome: AUC From Time Zero to Infinity (AUC[0-inf]) of Hydrochlorothiazide and Amiloride Hydrochloride in Plasma
Description: Blood samples were collected at indicated time points under fasting conditions for PK analysis of hydrochlorothiazide and amiloride. Bioequivalence of test product and reference product was assessed based on the 90 percent CIs for estimates of the geometric mean ratios between the AUC (0-inf) of the test and reference products in relation to the conventional bioequivalence range. An analysis of variance was used with sequence, subject (sequence), treatment and period as fixed effects. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 38 | 38
h*ng/mL
  Hydrochlorothiazide; n= 37, 38: number analyzed (Participants) | 37 | 38
  Hydrochlorothiazide; n= 37, 38 | 2310 (20.8) | 2490 (18.3)
  Amiloride; n= 22, 22: number analyzed (Participants) | 22 | 22
  Amiloride; n= 22, 22 | 117 (19.5) | 112 (18.2)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — Bioequivalence of hydrochlorothiazide and amiloride hydrochloride was determined; Least square mean ratio = 92.37, 90% CI 2-sided [88.75 to 96.12] — Comparison of Tmax of hydrochlorothiazide for test and reference product has been presented
Statistical Analysis 2: Comparison: Treatment A vs Treatment B; Test type: Other; Least square mean ratio = 101.47, 90% CI 2-sided [97.84 to 105.23] — Comparison of Tmax of amiloride for test and reference product has been presented

4. Secondary Outcome: Time of Occurrence of Cmax (Tmax) of Hydrochlorothiazide and Amiloride Hydrochloride in Plasma
Description: Blood samples were collected at indicated time points under fasting conditions for PK analysis of hydrochlorothiazide and amiloride. Median and full range has been presented.
Time Frame: as for outcome 1
Population: PK Population
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 38 | 38
Hour
  Hydrochlorothiazide | 2.505 [1.01 to 4.51] | 1.509 [0.67 to 3.50]
  Amiloride | 2.507 [1.50 to 4.51] | 2.508 [1.00 to 4.51]

5. Secondary Outcome: Percentage of AUC(0-inf) Obtained by Extrapolation (Percent AUCex) of Hydrochlorothiazide and Amiloride Hydrochloride in Plasma
Description: Blood samples were collected at indicated time points under fasting conditions for PK analysis of hydrochlorothiazide and amiloride. Bioequivalence of test product and reference product was assessed based on the 90 percent CIs for estimates of the geometric mean ratios between percent AUCex of the test and reference products in relation to the conventional bioequivalence range. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent of area
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 38 | 38
Percent of area
  Hydrochlorothiazide; n= 37, 38: number analyzed (Participants) | 37 | 38
  Hydrochlorothiazide; n= 37, 38 | 5.24 (37.7) | 4.63 (33.2)
  Amiloride; n= 22, 22: number analyzed (Participants) | 22 | 22
  Amiloride; n= 22, 22 | 9.68 (35.7) | 10.7 (44.9)

6. Secondary Outcome: Terminal Phase Half-life (T1/2) of Hydrochlorothiazide and Amiloride Hydrochloride in Plasma
Description: Blood samples were collected at indicated time points under fasting conditions for PK analysis of hydrochlorothiazide and amiloride. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: as for outcome 1
Population: PK Population
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 38 | 38
Hour
  Hydrochlorothiazide; n= 37, 38: number analyzed (Participants) | 37 | 38
  Hydrochlorothiazide; n= 37, 38 | 12.4 [8.47 to 18.8] | 11.3 [8.01 to 15.0]
  Amiloride; n= 22, 22: number analyzed (Participants) | 22 | 22
  Amiloride; n= 22, 22 | 15.2 [11.3 to 22.2] | 16.6 [10.9 to 23.8]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) During Treatment Period
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth effect, other situations and is associated with liver injury or impaired liver function. Only those participants with data available at the specified time points were analyzed
Time Frame: Up to 25 days
Population: Safety Population comprised of all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 40 | 40
Participants
  AEs | 5 | 8
  SAEs | 0 | 0

8. Secondary Outcome: Alanine Aminotransferase (ALT), Alkaline Phosphatase (Alk.Phosph.) and Aspartate Aminotransferase (AST) Levels at Indicated Time Points
Description: Serum ALT, alk. phosph. and AST levels were assessed as a clinical chemistry laboratory parameter at Day -1 and Day 3 in each treatment period. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Day -1 and Day 3 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Unit per liter (U/L)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 42 | 42
Unit per liter (U/L)
  ALT;Period 1 (P1);Day -1;24 hour pre-dose;n=21,21: number analyzed (Participants) | 21 | 21
  ALT;Period 1 (P1);Day -1;24 hour pre-dose;n=21,21 | 19.8 (10.55) | 16.6 (6.98)
  ALT; P1; Day 3; 48 hour post-dose; n= 21,20: number analyzed (Participants) | 21 | 20
  ALT; P1; Day 3; 48 hour post-dose; n= 21,20 | 15.9 (7.92) | 14.1 (5.49)
  ALT; P2; Day -1; 24 hour pre-dose; n= 19,19: number analyzed (Participants) | 19 | 19
  ALT; P2; Day -1; 24 hour pre-dose; n= 19,19 | 15.8 (7.03) | 17.6 (9.08)
  ALT; P2; Day 3; 48 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  ALT; P2; Day 3; 48 hour post-dose; n= 19, 19 | 15.8 (7.18) | 16.9 (10.00)
  Alk.phosph.; P1; Day -1; 24 hour pre-dose; n=21,21: number analyzed (Participants) | 21 | 21
  Alk.phosph.; P1; Day -1; 24 hour pre-dose; n=21,21 | 67.5 (16.59) | 71.1 (13.20)
  Alk.phosph.; P1; Day 3; 48 hour post-dose; n=21,20: number analyzed (Participants) | 21 | 20
  Alk.phosph.; P1; Day 3; 48 hour post-dose; n=21,20 | 67.1 (17.83) | 69.9 (14.06)
  Alk.phosph.; P2; Day -1; 24 hour pre-dose; n=19,19: number analyzed (Participants) | 19 | 19
  Alk.phosph.; P2; Day -1; 24 hour pre-dose; n=19,19 | 65.1 (12.52) | 63.6 (18.27)
  Alk.phosph.; P2; Day 3; 48 hour post-dose; n=19,19: number analyzed (Participants) | 19 | 19
  Alk.phosph.; P2; Day 3; 48 hour post-dose; n=19,19 | 66.8 (13.76) | 65.2 (15.66)
  AST; P1; Day -1; 24 hour pre-dose; n=21, 21: number analyzed (Participants) | 21 | 21
  AST; P1; Day -1; 24 hour pre-dose; n=21, 21 | 21.9 (8.56) | 20.1 (4.43)
  AST; P1; Day 3; 48 hour post-dose; n=21, 20: number analyzed (Participants) | 21 | 20
  AST; P1; Day 3; 48 hour post-dose; n=21, 20 | 17.5 (4.26) | 17.8 (3.81)
  AST; P2; Day -1; 24 hour pre-dose; n=19, 19: number analyzed (Participants) | 19 | 19
  AST; P2; Day -1; 24 hour pre-dose; n=19, 19 | 21.6 (5.81) | 21.1 (5.66)
  AST; P2; Day 3; 48 hour post-dose; n=19, 19: number analyzed (Participants) | 19 | 19
  AST; P2; Day 3; 48 hour post-dose; n=19, 19 | 19.9 (4.67) | 18.4 (5.67)

9. Secondary Outcome: Blood Urea Nitrogen (BUN) Levels at Indicated Time Points
Description: Serum BUN levels were assessed as a clinical chemistry laboratory parameter at Day -1 and Day 3 in each treatment period. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Day -1 and Day 3 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 42 | 42
Milligrams per deciliter (mg/dL)
  P1; Day-1; 24 hour pre-dose; n=21, 21: number analyzed (Participants) | 21 | 21
  P1; Day-1; 24 hour pre-dose; n=21, 21 | 12.519 (3.327) | 12.702 (3.954)
  P1; Day 3; 48 hour post-dose; n=21, 20: number analyzed (Participants) | 21 | 20
  P1; Day 3; 48 hour post-dose; n=21, 20 | 14.970 (3.626) | 15.593 (3.020)
  P2; Day -1; 24 hour pre-dose; n=19, 19: number analyzed (Participants) | 19 | 19
  P2; Day -1; 24 hour pre-dose; n=19, 19 | 12.185 (2.345) | 12.164 (3.216)
  P2; Day 3; 48 hour post-dose; n=19, 19: number analyzed (Participants) | 19 | 19
  P2; Day 3; 48 hour post-dose; n=19, 19 | 16.372 (4.446) | 15.208 (3.493)

10. Secondary Outcome: Calcium, Chloride, Glucose, Magnesium, Potassium and Sodium Levels at Indicated Time Points
Description: Serum calcium, chloride, glucose, magnesium, potassium and sodium levels were assessed as a clinical chemistry laboratory parameter at Day -1 and Day 3 in each treatment period. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Day -1 and Day 3 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter (Mmol/L)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 42 | 42
Millimoles per liter (Mmol/L)
  Calcium; P1; Day-1; 24 hour pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  Calcium; P1; Day-1; 24 hour pre-dose; n= 21, 21 | 2.400 (0.075) | 2.418 (0.085)
  Calcium; P1; Day 3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  Calcium; P1; Day 3; 48 hour post-dose; n= 21, 20 | 2.396 (0.078) | 2.393 (0.071)
  Calcium; P2; Day-1; 24 hour pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Calcium; P2; Day-1; 24 hour pre-dose; n= 19, 19 | 2.374 (0.053) | 2.335 (0.074)
  Calcium; P2; Day 3; 48 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Calcium; P2; Day 3; 48 hour post-dose; n= 19, 19 | 2.415 (0.078) | 2.379 (0.069)
  Chloride; P1; Day-1; 24 hour pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  Chloride; P1; Day-1; 24 hour pre-dose; n= 21, 21 | 104.80 (2.286) | 103.62 (2.225)
  Chloride; P1; Day 3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  Chloride; P1; Day 3; 48 hour post-dose; n= 21, 20 | 103.27 (1.755) | 102.63 (2.011)
  Chloride; P2; Day-1; 24 hour pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Chloride; P2; Day-1; 24 hour pre-dose; n= 19, 19 | 104.36 (1.729) | 104.85 (2.252)
  Chloride; P2; Day 3; 48 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Chloride; P2; Day 3; 48 hour post-dose; n= 19, 19 | 102.62 (1.985) | 103.49 (1.882)
  Glucose; P1; Day-1; 24 hour pre-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  Glucose; P1; Day-1; 24 hour pre-dose; n= 21, 20 | 4.746 (0.777) | 4.643 (0.427)
  Glucose; P1; Day 3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  Glucose; P1; Day 3; 48 hour post-dose; n= 21, 20 | 5.006 (0.597) | 4.827 (0.368)
  Glucose; P2; Day-1; 24 hour pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Glucose; P2; Day-1; 24 hour pre-dose; n= 19, 19 | 4.754 (0.316) | 4.765 (0.354)
  Glucose; P2; Day 3; 48 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Glucose; P2; Day 3; 48 hour post-dose; n= 19, 19 | 4.652 (0.357) | 4.732 (0.282)
  Magnesium; P1; Day-1; 24 hour pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  Magnesium; P1; Day-1; 24 hour pre-dose; n= 21, 21 | 0.782 (0.066) | 0.801 (0.049)
  Magnesium; P1; Day 3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  Magnesium; P1; Day 3; 48 hour post-dose; n= 21, 20 | 0.781 (0.039) | 0.804 (0.044)
  Magnesium; P2; Day-1; 24 hour pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Magnesium; P2; Day-1; 24 hour pre-dose; n= 19, 19 | 0.826 (0.053) | 0.805 (0.053)
  Magnesium; P2; Day 3; 48 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Magnesium; P2; Day 3; 48 hour post-dose; n= 19, 19 | 0.821 (0.051) | 0.783 (0.052)
  Potassium; P1; Day-1; 24 hour pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  Potassium; P1; Day-1; 24 hour pre-dose; n= 21, 21 | 4.287 (0.347) | 4.294 (0.390)
  Potassium; P1; Day 3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  Potassium; P1; Day 3; 48 hour post-dose; n= 21, 20 | 4.303 (0.346) | 4.222 (0.438)
  Potassium; P2; Day-1; 24 hour pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Potassium; P2; Day-1; 24 hour pre-dose; n= 19, 19 | 4.300 (0.374) | 4.225 (0.289)
  Potassium; P2; Day 3; 48 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Potassium; P2; Day 3; 48 hour post-dose; n= 19, 19 | 4.364 (0.303) | 4.336 (0.288)
  Sodium; P1; Day-1; 24 hour pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  Sodium; P1; Day-1; 24 hour pre-dose; n= 21, 21 | 140.86 (2.242) | 140.67 (1.958)
  Sodium; P1; Day 3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  Sodium; P1; Day 3; 48 hour post-dose; n= 21, 20 | 138.90 (1.480) | 139.25 (1.410)
  Sodium; P2; Day-1; 24 hour pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Sodium; P2; Day-1; 24 hour pre-dose; n= 19, 19 | 140.11 (1.410) | 139.68 (2.187)
  Sodium; P2; Day 3; 48 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Sodium; P2; Day 3; 48 hour post-dose; n= 19, 19 | 139.11 (1.761) | 139.11 (2.424)

11. Secondary Outcome: Creatinine, Direct Bilirubin and Total Bilirubin Levels at Indicated Time Points
Description: Serum creatinine, direct bilirubin and total bilirubin levels were assessed as a clinical chemistry laboratory parameter at Day -1 and Day 3 in each treatment period. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Day -1 and Day 3 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 42 | 42
Micromoles per liter (µmol/L)
  Creatinine; P1; Day-1; 24 hour pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  Creatinine; P1; Day-1; 24 hour pre-dose; n= 21, 21 | 85.2 (13.69) | 85.0 (11.51)
  Creatinine; P1; Day3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  Creatinine; P1; Day3; 48 hour post-dose; n= 21, 20 | 87.0 (15.26) | 87.3 (12.18)
  Creatinine; P2; Day-1; 24 hour pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Creatinine; P2; Day-1; 24 hour pre-dose; n= 19, 19 | 82.1 (10.99) | 82.5 (13.33)
  Creatinine; P2; Day3; 48 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  Creatinine; P2; Day3; 48 hour post-dose; n= 19, 19 | 85.6 (15.31) | 88.7 (16.69)
  Direct bilirubin;P1;Day-1;24 hour pre-dose;n=21,21: number analyzed (Participants) | 21 | 21
  Direct bilirubin;P1;Day-1;24 hour pre-dose;n=21,21 | 4.25 (1.771) | 4.52 (1.825)
  Direct bilirubin;P1;Day3;48 hour post-dose;n=21,20: number analyzed (Participants) | 21 | 20
  Direct bilirubin;P1;Day3;48 hour post-dose;n=21,20 | 3.20 (1.599) | 3.72 (1.493)
  Direct bilirubin;P2;Day-1;24 hour pre-dose;n=19,19: number analyzed (Participants) | 19 | 19
  Direct bilirubin;P2;Day-1;24 hour pre-dose;n=19,19 | 3.94 (1.357) | 3.64 (1.446)
  Direct bilirubin;P2;Day3;48 hour post-dose;n=19,19: number analyzed (Participants) | 19 | 19
  Direct bilirubin;P2;Day3;48 hour post-dose;n=19,19 | 3.77 (1.559) | 3.14 (1.340)
  Total bilirubin;P1;Day-1;24 hour pre-dose;n=21,21: number analyzed (Participants) | 21 | 21
  Total bilirubin;P1;Day-1;24 hour pre-dose;n=21,21 | 12.10 (6.208) | 13.48 (6.923)
  Total bilirubin;P1;Day3;48 hour post-dose;n=21,20: number analyzed (Participants) | 21 | 20
  Total bilirubin;P1;Day3;48 hour post-dose;n=21,20 | 9.40 (5.265) | 10.80 (5.601)
  Total bilirubin;P2;Day-1;24 hour pre-dose;n=19,19: number analyzed (Participants) | 19 | 19
  Total bilirubin;P2;Day-1;24 hour pre-dose;n=19,19 | 10.61 (4.651) | 10.08 (5.119)
  Total bilirubin;P2;Day3;48 hour post-dose;n=19,19: number analyzed (Participants) | 19 | 19
  Total bilirubin;P2;Day3;48 hour post-dose;n=19,19 | 10.83 (5.920) | 8.67 (4.492)

12. Secondary Outcome: Total Protein Levels at Indicated Time Points
Description: Serum total protein levels were assessed as a clinical chemistry laboratory parameter at Day -1 and Day 3 in each treatment period. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Day -1 and Day 3 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 42 | 42
Grams per liter (g/L)
  P1; Day-1; 24 hours pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day-1; 24 hours pre-dose; n= 21, 21 | 74.08 (4.943) | 76.06 (3.733)
  P1; Day 3; 48 hours post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  P1; Day 3; 48 hours post-dose; n= 21, 20 | 74.53 (5.259) | 74.99 (3.844)
  P2; Day-1; 24 hours pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day-1; 24 hours pre-dose; n= 19, 19 | 71.29 (3.369) | 70.06 (4.002)
  P2; Day 3; 48 hours post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day 3; 48 hours post-dose; n= 19, 19 | 73.56 (3.676) | 72.33 (4.241)

13. Secondary Outcome: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Values at Indicated Time Points
Description: Vital sign measurements including SBP and DBP were taken in a supine position after at least 5 minutes of rest at Day -1, Day 1, Day 2 and Day 3 in each treatment period. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1 and Day 3 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 42 | 42
Millimeters of mercury (mmHg)
  SBP; P1; Day-1; 12 hour pre-dose; n=21,21: number analyzed (Participants) | 21 | 21
  SBP; P1; Day-1; 12 hour pre-dose; n=21,21 | 115.9 (6.88) | 115.8 (8.99)
  SBP; P1; Day1; 1 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  SBP; P1; Day1; 1 hour post-dose; n= 21, 21 | 112.8 (8.90) | 111.6 (7.56)
  SBP; P1; Day1; 1.5 hour pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  SBP; P1; Day1; 1.5 hour pre-dose; n= 21, 21 | 111.5 (8.15) | 110.8 (11.01)
  SBP; P1; Day1; 2 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  SBP; P1; Day1; 2 hour post-dose; n= 21, 21 | 113.3 (9.59) | 112.6 (7.95)
  SBP: P1; Day1; 4 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  SBP: P1; Day1; 4 hour post-dose; n= 21, 21 | 112.5 (8.66) | 114.0 (9.30)
  SBP; P1; Day1; 6 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  SBP; P1; Day1; 6 hour post-dose; n= 21, 21 | 110.9 (6.69) | 113.0 (8.26)
  SBP; P1; Day1; 8 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  SBP; P1; Day1; 8 hour post-dose; n= 21, 21 | 113.0 (8.66) | 111.8 (8.62)
  SBP; P1; Day2; 24 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  SBP; P1; Day2; 24 hour post-dose; n= 21, 21 | 111.4 (6.99) | 110.5 (6.79)
  SBP; P1; Day3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  SBP; P1; Day3; 48 hour post-dose; n= 21, 20 | 114.5 (9.11) | 113.8 (9.20)
  SBP; P2; Day-1; 12 hour pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  SBP; P2; Day-1; 12 hour pre-dose; n= 19, 19 | 113.8 (7.38) | 116.2 (10.04)
  SBP; P2; Day1; 1 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  SBP; P2; Day1; 1 hour post-dose; n= 19, 19 | 110.0 (8.54) | 113.7 (11.71)
  SBP; P2; Day1; 1.5 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  SBP; P2; Day1; 1.5 hour post-dose; n= 19, 19 | 108.9 (8.14) | 112.2 (12.62)
  SBP; P2; Day1; 2 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  SBP; P2; Day1; 2 hour post-dose; n= 19, 19 | 109.6 (7.73) | 113.8 (12.49)
  SBP: P2; Day1; 4 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  SBP: P2; Day1; 4 hour post-dose; n= 19, 19 | 109.5 (9.54) | 113.5 (11.57)
  SBP: P2; Day1; 6 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  SBP: P2; Day1; 6 hour post-dose; n= 19, 19 | 108.5 (7.57) | 112.4 (10.79)
  SBP: P2; Day1; 8 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  SBP: P2; Day1; 8 hour post-dose; n= 19, 19 | 109.8 (8.53) | 111.5 (12.04)
  SBP: P2; Day2; 24 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  SBP: P2; Day2; 24 hour post-dose; n= 19, 19 | 109.1 (7.13) | 110.6 (10.03)
  SBP; P2; Day3; 48 hour post-dose; n= 18, 19: number analyzed (Participants) | 18 | 19
  SBP; P2; Day3; 48 hour post-dose; n= 18, 19 | 112.9 (8.56) | 116.5 (9.18)
  DBP; P1; Day-1; 12 hour pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  DBP; P1; Day-1; 12 hour pre-dose; n= 21, 21 | 65.4 (7.32) | 64.9 (7.25)
  DBP; P1; Day1; 1 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  DBP; P1; Day1; 1 hour post-dose; n= 21, 21 | 63.7 (6.79) | 63.5 (5.55)
  DBP: P1; Day1; 1.5 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  DBP: P1; Day1; 1.5 hour post-dose; n= 21, 21 | 64.0 (7.08) | 63.9 (8.57)
  DBP; P1; Day1; 2 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  DBP; P1; Day1; 2 hour post-dose; n= 21, 21 | 63.4 (7.10) | 65.7 (9.45)
  DBP: P1; Day1; 4 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  DBP: P1; Day1; 4 hour post-dose; n= 21, 21 | 64.8 (6.82) | 64.4 (7.21)
  DBP; P1; Day1; 6 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  DBP; P1; Day1; 6 hour post-dose; n= 21, 21 | 61.4 (4.34) | 62.7 (6.20)
  DBP; P1; Day1; 8 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  DBP; P1; Day1; 8 hour post-dose; n= 21, 21 | 63.0 (6.00) | 63.7 (6.02)
  DBP: P1; Day2; 24 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  DBP: P1; Day2; 24 hour post-dose; n= 21, 21 | 64.9 (5.06) | 64.2 (5.86)
  DBP: P1; Day3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  DBP: P1; Day3; 48 hour post-dose; n= 21, 20 | 67.3 (5.55) | 66.0 (6.38)
  DBP; P2; Day-1; 12 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  DBP; P2; Day-1; 12 hour post-dose; n= 19, 19 | 63.1 (6.03) | 65.8 (7.65)
  DBP; P2; Day1; 1 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  DBP; P2; Day1; 1 hour post-dose; n= 19, 19 | 63.9 (6.86) | 64.1 (8.39)
  DBP; P2; Day1; 1.5 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  DBP; P2; Day1; 1.5 hour post-dose; n= 19, 19 | 61.1 (5.36) | 63.4 (8.64)
  DBP; P2; Day1; 2 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  DBP; P2; Day1; 2 hour post-dose; n= 19, 19 | 62.5 (6.87) | 65.3 (7.28)
  DBP; P2; Day1; 4 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  DBP; P2; Day1; 4 hour post-dose; n= 19, 19 | 62.8 (7.73) | 65.3 (8.08)
  DBP: P2; Day1; 6 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  DBP: P2; Day1; 6 hour post-dose; n= 19, 19 | 59.4 (5.85) | 61.5 (6.33)
  DBP; P2; Day1; 8 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  DBP; P2; Day1; 8 hour post-dose; n= 19, 19 | 61.1 (5.91) | 62.9 (6.75)
  DBP: P2; Day2; 24 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  DBP: P2; Day2; 24 hour post-dose; n= 19, 19 | 62.9 (5.62) | 64.4 (7.79)
  DBP: P2; Day3; 48 hour post-dose; n= 18, 19: number analyzed (Participants) | 18 | 19
  DBP: P2; Day3; 48 hour post-dose; n= 18, 19 | 65.9 (7.28) | 67.2 (6.64)

14. Secondary Outcome: Respiratory Rate Values at Indicated Time Points
Description: Vital sign measurements including respiratory rate were taken in a supine position after at least 5 minutes of rest at Day -1, Day 1, Day 2 and Day 3 in each treatment period. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1 and Day 3 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 42 | 42
Breaths per minute
  P1; Day-1; 12 hour pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day-1; 12 hour pre-dose; n= 21, 21 | 16.5 (1.63) | 17.0 (1.45)
  P1; Day1; 1 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 1 hour post-dose; n= 21, 21 | 16.3 (2.70) | 17.0 (2.33)
  P1; Day1; 1.5 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 1.5 hour post-dose; n= 21, 21 | 16.7 (1.91) | 17.9 (1.62)
  P1; Day1; 2 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 2 hour post-dose; n= 21, 21 | 17.0 (2.06) | 17.5 (2.36)
  P1; Day1; 4 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 4 hour post-dose; n= 21, 21 | 16.9 (2.49) | 17.0 (2.25)
  P1; Day1; 6 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 6 hour post-dose; n= 21, 21 | 17.2 (2.49) | 18.4 (2.16)
  P1; Day1; 8 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 8 hour post-dose; n= 21, 21 | 16.9 (2.24) | 18.2 (1.89)
  P1; Day2; 24 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day2; 24 hour post-dose; n= 21, 21 | 18.2 (1.41) | 18.0 (1.80)
  P1; Day3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  P1; Day3; 48 hour post-dose; n= 21, 20 | 17.1 (1.53) | 17.7 (1.89)
  P2; Day-1; 12 hour pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day-1; 12 hour pre-dose; n= 19, 19 | 17.9 (1.47) | 17.2 (1.54)
  P2; Day1; 1 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 1 hour post-dose; n= 19, 19 | 17.7 (2.03) | 17.9 (1.56)
  P2; Day1; 1.5 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 1.5 hour post-dose; n= 19, 19 | 15.8 (1.65) | 16.3 (1.82)
  P2; Day1; 2 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 2 hour post-dose; n= 19, 19 | 18.0 (1.89) | 17.3 (2.84)
  P2; Day1; 4 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 4 hour post-dose; n= 19, 19 | 17.9 (2.26) | 17.4 (2.50)
  P2; Day1; 6 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 6 hour post-dose; n= 19, 19 | 17.2 (1.92) | 18.3 (2.52)
  P2; Day1; 8 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 8 hour post-dose; n= 19, 19 | 18.7 (1.52) | 18.2 (2.10)
  P2; Day2; 24 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day2; 24 hour post-dose; n= 19, 19 | 17.5 (2.72) | 17.6 (1.64)
  P2; Day3; 48 hour post-dose; n= 18, 19: number analyzed (Participants) | 18 | 19
  P2; Day3; 48 hour post-dose; n= 18, 19 | 18.4 (1.62) | 17.2 (2.42)

15. Secondary Outcome: Pulse Rate Values at Indicated Time Points
Description: Vital sign measurements including pulse rate were taken in a supine position after at least 5 minutes of rest at Day -1, Day 1, Day 2 and Day 3 in each treatment period. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1 and Day 3 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 42 | 42
Beats per minute (bpm)
  P1; Day-1; 12 hour pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day-1; 12 hour pre-dose; n= 21, 21 | 66.9 (9.22) | 64.7 (9.57)
  P1; Day1; 1 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 1 hour post-dose; n= 21, 21 | 61.8 (11.26) | 62.0 (10.26)
  P1; Day1; 1.5 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 1.5 hour post-dose; n= 21, 21 | 62.5 (10.95) | 60.9 (11.05)
  P1; Day1; 2 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 2 hour post-dose; n= 21, 21 | 61.7 (10.55) | 60.7 (8.97)
  P1; Day1; 4 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 4 hour post-dose; n= 21, 21 | 64.1 (11.32) | 62.5 (9.91)
  P1; Day1; 6 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 6 hour post-dose; n= 21, 21 | 71.5 (13.85) | 70.8 (10.17)
  P1; Day1; 8 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 8 hour post-dose; n= 21, 21 | 66.0 (9.93) | 67.8 (9.33)
  P1; Day2; 24 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day2; 24 hour post-dose; n= 21, 21 | 69.0 (11.26) | 68.6 (10.18)
  P1; Day3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  P1; Day3; 48 hour post-dose; n= 21, 20 | 71.4 (12.93) | 73.0 (9.49)
  P2; Day-1; 12 hour pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day-1; 12 hour pre-dose; n= 19, 19 | 65.2 (9.15) | 65.2 (11.95)
  P2; Day1; 1 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 1 hour post-dose; n= 19, 19 | 62.5 (8.82) | 60.1 (9.72)
  P2; Day1; 1.5 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 1.5 hour post-dose; n= 19, 19 | 61.5 (8.02) | 62.8 (10.97)
  P2; Day1; 2 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 2 hour post-dose; n= 19, 19 | 60.7 (8.33) | 59.2 (8.60)
  P2; Day1; 4 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 4 hour post-dose; n= 19, 19 | 62.4 (8.58) | 62.7 (11.36)
  P2; Day1; 6 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 6 hour post-dose; n= 19, 19 | 72.9 (8.23) | 71.4 (13.25)
  P2; Day1; 8 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 8 hour post-dose; n= 19, 19 | 68.2 (8.89) | 66.2 (11.26)
  P2; Day2; 24 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day2; 24 hour post-dose; n= 19, 19 | 69.0 (9.99) | 68.8 (13.29)
  P2; Day3; 48 hour post-dose; n= 18, 19: number analyzed (Participants) | 18 | 19
  P2; Day3; 48 hour post-dose; n= 18, 19 | 70.3 (11.69) | 73.4 (17.13)

16. Secondary Outcome: Body Temperature Values at Indicated Time Points
Description: Vital sign measurements including body temperature were taken in a supine position after at least 5 minutes of rest at Day -1, Day 1, Day 2 and Day 3 in each treatment period. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Day -1 and Day 3 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 42 | 42
Degree Celsius
  P1; Day-1; 12 hour pre-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day-1; 12 hour pre-dose; n= 21, 21 | 36.42 (0.339) | 36.43 (0.376)
  P1; Day1; 1 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 1 hour post-dose; n= 21, 21 | 36.44 (0.262) | 36.40 (0.392)
  P1; Day1; 1.5 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 1.5 hour post-dose; n= 21, 21 | 36.06 (0.294) | 36.05 (0.314)
  P1; Day1; 2 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 2 hour post-dose; n= 21, 21 | 36.42 (0.339) | 36.38 (0.314)
  P1; Day1; 4 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 4 hour post-dose; n= 21, 21 | 36.45 (0.364) | 36.46 (0.365)
  P1; Day1; 6 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 6 hour post-dose; n= 21, 21 | 36.59 (0.422) | 36.61 (0.309)
  P1; Day1; 8 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day1; 8 hour post-dose; n= 21, 21 | 36.64 (0.461) | 36.75 (0.357)
  P1; Day2; 24 hour post-dose; n= 21, 21: number analyzed (Participants) | 21 | 21
  P1; Day2; 24 hour post-dose; n= 21, 21 | 36.28 (0.387) | 36.30 (0.322)
  P1; Day3; 48 hour post-dose; n= 21, 20: number analyzed (Participants) | 21 | 20
  P1; Day3; 48 hour post-dose; n= 21, 20 | 36.26 (0.334) | 36.28 (0.374)
  P2; Day-1; 12 hour pre-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day-1; 12 hour pre-dose; n= 19, 19 | 36.41 (0.358) | 36.34 (0.383)
  P2; Day1; 1 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 1 hour post-dose; n= 19, 19 | 36.28 (0.302) | 36.24 (0.435)
  P2; Day1; 1.5 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 1.5 hour post-dose; n= 19, 19 | 36.06 (0.263) | 36.19 (0.336)
  P2; Day1; 2 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 2 hour post-dose; n= 19, 19 | 36.41 (0.294) | 36.38 (0.405)
  P2; Day1; 4 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 4 hour post-dose; n= 19, 19 | 36.53 (0.335) | 36.44 (0.380)
  P2; Day1; 6 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 6 hour post-dose; n= 19, 19 | 36.59 (0.331) | 36.57 (0.406)
  P2; Day1; 8 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day1; 8 hour post-dose; n= 19, 19 | 36.64 (0.383) | 36.65 (0.399)
  P2; Day2; 24 hour post-dose; n= 19, 19: number analyzed (Participants) | 19 | 19
  P2; Day2; 24 hour post-dose; n= 19, 19 | 36.15 (0.301) | 36.17 (0.437)
  P2; Day3; 48 hour post-dose; n= 18, 19: number analyzed (Participants) | 18 | 19
  P2; Day3; 48 hour post-dose; n= 18, 19 | 36.08 (0.323) | 36.28 (0.486)

ADVERSE EVENTS:
Time Frame: On-therapy serious adverse events (SAEs) and non-serious AEs are presented from the start of study treatment up to follow up visit 7 days post-last dose (Up to 25 days).
Description: On-therapy SAEs and non-serious AEs are reported for the safety Population, comprising of all participants who received at least one dose of study treatment.
Arm/Group | Treatment A | Treatment B
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 5/40 | 13/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=40) | Treatment B (N=40)
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Crystal Urine (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 5
Headache (Nervous system disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT03031496/Prot_SAP_000.pdf